CLINICAL TRIAL: NCT05498909
Title: A Real-world Registry Study of Multidisciplinary Collaborative Diagnosis and Treatment Model for Cardioembolic Stroke
Acronym: CSMDT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Xiao Huang (Other)
Responsible Party: Sponsor-Investigator, Xiao Huang, Principal Investigator, Second Affiliated Hospital of Nanchang University
Organization: Second Affiliated Hospital of Nanchang University (Other)
Other Study IDs: 2022-01
Record Dates: First submitted 2022-08-08; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Cardioembolic Stroke; Multidisciplinary Communication
Keywords: Cardioembolic stroke; MDT; atrial fibrillation; Valvular heart disease; PFO
MeSH Terms: conditions — Embolic Stroke; Atrial Fibrillation; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Collect blood samples, tissues and body fluids according to the requirements of the sample bank
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Treatment group: Treatment group（Multidisciplinary assisted treatment model group）： Those who received any of the following treatments, as recommended by the standard medical procedure, were considered to have received the standard medical treatment; otherwise, they were not.
  1. Surgical procedures: left atrial appendage ligation, left atrial appendage clip, valve repair or replacement, etc.
  2. Medical procedures: atrial fibrillation radiofrequency ablation, valvular closure, left atrial appendage closure, etc.
  3. Anticoagulant drug therapy: standardized anticoagulant drug therapy.
  Interventions: Other: Multidisciplinary joint diagnosis and treatment mode
- Control group: Control group（Routine diagnosis and treatment model group）:
  Patients who did not agree to enter the multidisciplinary treatment mode were automatically admitted to the routine treatment mode group

INTERVENTIONS:
Other: Multidisciplinary joint diagnosis and treatment mode — Multidisciplinary joint diagnosis and treatment mode,break down barriers and treat the heart and brain together
  Groups: Treatment group

SUMMARY:
Study Title: A real-world registry of multidisciplinary collaborative diagnosis and treatment models for cardioembolic stroke

Research Objectives:

① Main objective: To establish a multidisciplinary assisted diagnosis and treatment model for patients at high risk of cardioembolic stroke, manage and collect the diagnosis, treatment and prognosis data of patients.

② Secondary objective: To investigate the improvement of cardioembolic stroke, cardiovascular complex events, recurrent stroke and all-cause mortality risk, quality of life, and cardiac function between the "multidisciplinary assisted treatment model" group and the "conventional treatment model group". The routine diagnosis and treatment mode can match the patients who did not adopt the "multidisciplinary assisted diagnosis and treatment mode" in the same period.

Type of design: A prospective, observational, real-world study. No fixed diagnosis and treatment plan was established in advance, and only a multidisciplinary assisted diagnosis and treatment model was established. All treatment choices were made by clinicians according to the expert consensus of relevant textbooks and clinical guidelines, and according to the patient's condition.

Subjects: From September 2022 to September 2023, high-risk patients with cardioembolic stroke were collected from the Second Affiliated Hospital of Nanchang University and sub-centers of hospitals at all levels in Jiangxi Province.

DETAILED DESCRIPTION:
Summary of Research Protocol:

Study Title: A real-world registry of multidisciplinary collaborative diagnosis and treatment models for cardioembolic stroke

Research Objectives:

① Main objective: To establish a multidisciplinary assisted diagnosis and treatment model for patients at high risk of cardioembolic stroke, manage and collect the diagnosis, treatment and prognosis data of patients.

② Secondary objective: To investigate the improvement of cardioembolic stroke, cardiovascular complex events, recurrent stroke and all-cause mortality risk, quality of life, and cardiac function between the "multidisciplinary assisted treatment model" group and the "conventional treatment model group". The routine diagnosis and treatment mode can match the patients who did not adopt the "multidisciplinary assisted diagnosis and treatment mode" in the same period.

Type of design: A prospective, observational, real-world study. No fixed diagnosis and treatment plan was established in advance, and only a multidisciplinary assisted diagnosis and treatment model was established. All treatment choices were made by clinicians according to the expert consensus of relevant textbooks and clinical guidelines, and according to the patient's condition.

Subjects: From September 2022 to September 2023, high-risk patients with cardioembolic stroke were collected from the Second Affiliated Hospital of Nanchang University and sub-centers of hospitals at all levels in Jiangxi Province.

Multidisciplinary assisted care mode group: Patients who agreed to and accepted the recommendation of multidisciplinary assisted care mode were enrolled in the multidisciplinary assisted care mode group. These patients would undergo further stroke (primary/secondary) prevention intervention.

Those who received any of the following treatments, as recommended by the standard medical procedure, were considered to have received the standard medical treatment; otherwise, they were not.

1. Surgical procedures: left atrial appendage ligation, left atrial appendage clip, valve repair or replacement, etc.
2. Medical procedures: atrial fibrillation radiofrequency ablation, valvular closure, left atrial appendage closure, etc.
3. Anticoagulant drug therapy: standardized anticoagulant drug therapy.

Routine treatment mode group: Patients who did not agree to enter the multidisciplinary treatment mode were automatically entered into the routine treatment mode group.

ELIGIBILITY:
Inclusion Criteria:

* The risk of high embolism (including intracardiac thrombosis, intracardiac tumor, aortic atherosclerosis, atrial fibrillation and spontaneous ultrasound imaging) was in line with the risk stratification criteria of Chinese Expert Consensus on the Diagnosis of cardiogenic Stroke (2020);
* In accordance with the Chinese Expert Consensus on the Treatment of cardiogenic Stroke (2022), surgical indications for cardiac diseases (including left atrial appendage closure, left atrial appendage ligation, and radiofrequency ablation of atrial fibrillation are recommended for high-risk stroke patients with atrial fibrillation; For cryptogenic stroke patients with high-risk PFO, transcatheter PFO closure is recommended. Valve repair or replacement);
* Understand and voluntarily sign the informed consent.

Exclusion Criteria:

* Serious mental disorder, unable to express the will;
* In the judgment of the investigator, there are obvious other abnormal signs, laboratory tests and clinical diseases, which are not suitable for investigator participation;
* Researchers judged that long-term follow-up could not be completed

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients at high risk of cardiogenic stroke in the Second Affiliated Hospital of Nanchang University and sub-centers of hospitals at all levels in Jiangxi Province from September 2022 to September 2023 were collected.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite end point of cardiovascular and cerebrovascular events | 1.5 years
  Non-fatal ischemic stroke, non-fatal hemorrhagic stroke, non-fatal myocardial infarction, non-fatal heart failure, cardiovascular and cerebrovascular death

SECONDARY OUTCOMES:
Cardiovascular and cerebrovascular death, All-cause death, Cardiac insufficiency, Cognitive dysfunction | 1.5 years
  Cardiovascular and cerebrovascular death, All-cause death, Cardiac insufficiency, Cognitive dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Xingen Zhu, President, Principal Investigator — Second Affiliated Hospital of Nanchang University
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lin SP, Long Y, Chen XH, Lin PY, Jiang HL. STAF score is a new simple approach for diagnosing cardioembolic stroke. Int J Neurosci. 2017 Mar;127(3):261-266. doi: 10.1080/00207454.2016.1185715. Epub 2016 May 25. PMID 27211997
- [Result] Marnane M, Duggan CA, Sheehan OC, Merwick A, Hannon N, Curtin D, Harris D, Williams EB, Horgan G, Kyne L, McCormack PM, Duggan J, Moore A, Crispino-O'Connell G, Kelly PJ. Stroke subtype classification to mechanism-specific and undetermined categories by TOAST, A-S-C-O, and causative classification system: direct comparison in the North Dublin population stroke study. Stroke. 2010 Aug;41(8):1579-86. doi: 10.1161/STROKEAHA.109.575373. Epub 2010 Jul 1. PMID 20595675
- [Result] Vahanian A, Alfieri O, Andreotti F, Antunes MJ, Baron-Esquivias G, Baumgartner H, Borger MA, Carrel TP, De Bonis M, Evangelista A, Falk V, Lung B, Lancellotti P, Pierard L, Price S, Schafers HJ, Schuler G, Stepinska J, Swedberg K, Takkenberg J, Von Oppell UO, Windecker S, Zamorano JL, Zembala M; ESC Committee for Practice Guidelines (CPG); Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC); European Association for Cardio-Thoracic Surgery (EACTS). Guidelines on the management of valvular heart disease (version 2012): the Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS). Eur J Cardiothorac Surg. 2012 Oct;42(4):S1-44. doi: 10.1093/ejcts/ezs455. Epub 2012 Aug 25. No abstract available. PMID 22922698
- [Result] Friedman DJ, Piccini JP, Wang T, Zheng J, Malaisrie SC, Holmes DR, Suri RM, Mack MJ, Badhwar V, Jacobs JP, Gaca JG, Chow SC, Peterson ED, Brennan JM. Association Between Left Atrial Appendage Occlusion and Readmission for Thromboembolism Among Patients With Atrial Fibrillation Undergoing Concomitant Cardiac Surgery. JAMA. 2018 Jan 23;319(4):365-374. doi: 10.1001/jama.2017.20125. PMID 29362794
- [Result] Lee PH, Song JK, Kim JS, Heo R, Lee S, Kim DH, Song JM, Kang DH, Kwon SU, Kang DW, Lee D, Kwon HS, Yun SC, Sun BJ, Park JH, Lee JH, Jeong HS, Song HJ, Kim J, Park SJ. Cryptogenic Stroke and High-Risk Patent Foramen Ovale: The DEFENSE-PFO Trial. J Am Coll Cardiol. 2018 May 22;71(20):2335-2342. doi: 10.1016/j.jacc.2018.02.046. Epub 2018 Mar 12. PMID 29544871
- [Result] MacDougall NJ, Amarasinghe S, Muir KW. Secondary prevention of stroke. Expert Rev Cardiovasc Ther. 2009 Sep;7(9):1103-15. doi: 10.1586/erc.09.77. PMID 19764863
- [Result] Khoo CW, Lip GY. Clinical outcomes of acute stroke patients with atrial fibrillation. Expert Rev Cardiovasc Ther. 2009 Apr;7(4):371-4. doi: 10.1586/erc.09.11. PMID 19379061

DOCUMENTS (1):
  • Study Protocol (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT05498909/Prot_000.pdf